CLINICAL TRIAL: NCT00629538
Title: Effect of Therapeutic Thoracentesis on Cardiopulmonary Function in Patients With Congestive Heart Failure Complicated With Large to Massive Pleural Effusion
Brief Title: Therapeutic Thoracentesis for Patients With Congestive Heart Failure and Large Pleural Effusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Chung, Chi-Li/Chest physician of Department of Internal Medicine, Taipei Medical University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMUHIRB20070304
Record Dates: First submitted 2008-02-25; First posted 2008-03-06 (Estimated); Last update posted 2010-12-30 (Estimated); Status verified 2010-12

CONDITIONS: Congestive Heart Failure; Transudative Pleural Effusion
Keywords: congestive heart failure; thoracentesis; transudative pleural effusions
MeSH Terms: conditions — Heart Failure; Hydrothorax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Therapeutic thoracentesis — Thoracentesis was performed with drainage of 500 ml of pleural fluid first and every 200 ml thereafter until pleural pressure was lower than -20 cm H2O, chest discomfort developed, or no more pleural fluid could be removed.

SUMMARY:
Transudative pleural effusions are a common manifestation of patients with congestive heart failure. Severe dyspnea and respiratory failure may develop in those with large effusions, which in general show poor response to medical treatment. Therapeutic thoracenteses (TT) may be indicated in these patients and can produce marked relief of symptoms. However, the underlying effect of TT on gas exchange and respiratory mechanics in theses patients remains unclear. The researchers' hypothesis is that,TT may improve arterial oxygenation and respiratory mechanics in patients with congestive heart failure complicated by large pleural effusions.

ELIGIBILITY:
Inclusion Criteria:

* transudative pleural effusion established by the criteria of Light
* the effusion occupying at least half of one hemithorax shown on chest radiography
* symptoms of respiratory distress
* diagnosis of congestive heart failure

Exclusion Criteria:

* severe uncontrolled coagulopathy
* unstable hemodynamics
* diagnosis of liver cirrhosis, chronic obstructive pulmonary disease,asthma and/or any parenchymal lung disease, such as pneumonia, fibrosis or malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Vital signs, minute volume, expiratory tidal volume, dynamic compliance, arterial oxygen saturation and arterial blood gases, the volume of pleural fluid removed, and the changes in pleural liquid pressure and pleural space elastance | 15 minutes after therapeutic thoracentesis

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Li Chung, MD, PhD, Principal Investigator — Department of Internal Medicine, Taipei Medical University Hospital
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chen WL, Chung CL, Hsiao SH, Chang SC. Pleural space elastance and changes in oxygenation after therapeutic thoracentesis in ventilated patients with heart failure and transudative pleural effusions. Respirology. 2010 Aug;15(6):1001-8. doi: 10.1111/j.1440-1843.2010.01812.x. Epub 2010 Jul 20. PMID 20646242